CLINICAL TRIAL: NCT02537418
Title: A Phase IB Study of Durvalumab (MEDI4736) With or Without Tremelimumab in Patients With Advanced Incurable Solid Malignancies Given With or Without Standard Chemotherapy Regimens
Brief Title: Durvalumab With or Without Tremelimumab in Advanced Incurable Solid Malignancies Given With or Without Standard Chemotherapy Regimens
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: I226
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Solid Malignancies
MeSH Terms: interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- durvalumab ± tremelimumab (Experimental): durvalumab; Day 1 every 3 weeks or 4 weeks
  tremelimumab; every 3-6 weeks for a total of 1-6 doses
  Interventions: Drug: durvalumab; Drug: tremelimumab

INTERVENTIONS:
Drug: durvalumab
Drug: tremelimumab

SUMMARY:
The purpose of this study is to find the highest dose of durvalumab or of durvalumab with tremelimumab that can be tolerated without causing very severe side effects when receiving standard chemotherapy and to see what effects the study drugs has on this type of cancer. Patients may receive durvalumab alone or in combination with tremelimumab.

DETAILED DESCRIPTION:
The researchers doing this study are also interested in looking for markers that will help predict which patients are most likely to be helped by the study drugs, durvalumab and tremelimumab. This is done by starting at a dose lower than the one that does not cause side effects in animals. Participants are given durvalumab alone or durvalumab together with tremelimumab and are watched very closely to see what side effects they have and to make sure the side effects are not severe. If the side effects are not severe, then new participants will be given a higher dose of durvalumab together with tremelimumab. Participants joining this study later on will get higher doses of durvalumab together with tremelimumab than participants who join earlier. This will continue until a dose is found that causes severe but temporary side effects. Doses higher than that will not be given.

The second purpose is to see if there are any differences in the side effects and the way durvalumab and tremelimumab are handled in your body when durvalumab is given together at the same time with tremelimumab compared to when durvalumab is given after tremelimumab. This is called dose level five.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically and/or cytologically confirmed cancer that is advanced / metastatic / recurrent or unresectable and for which no curative therapy exists.

  * Patients must be considered suitable candidates for and eligible to receive one of the regimens (including durvalumab and tremelimumab alone (dose level 5) included in this protocol and which is open to accrual. For each regimen, specific criteria for registration may be applicable to the cohort/dose level to ensure tolerability in the planned phase II or III trials. Centres must confirm that the planned cohort is open to accrual and whether there are any restrictions on tumour types prior to approaching patients.
  * For etoposide/carboplatin regimen, patients must have untreated small cell lung cancer (SCLC).
  * If a formalin fixed paraffin embedded tissue block (from their primary or metastatic tumour) is available, patients must have provided informed consent for the release of the block. All patients must have provided informed consent for correlative studies.
  * Presence of clinically and/or radiologically documented disease. All radiology studies must be performed within 28 days prior to registration (within 35 days if negative). Patients ideally should have measurable disease.
  * Patients must have an ECOG performance status of 0, 1, or 2 (0 or 1 for untreated SCLC enrolled to etoposide/carboplatin). Patients with PS 2 must be considered fit for first line cytotoxic or immune based therapy and discussed with CCTG prior to enrolment.

Previous Therapy

• Cytotoxic Chemotherapy:

All Cohorts Except Etoposide-Carboplatin:

• Patients should not have received prior chemotherapy for advanced disease. Exceptions may be made for selected patients and regimens. Patients planned for dose level 5 may have received one line or prior chemotherapy. Consult CCTG before approaching patients.

Notes: Patients planned for cisplatin regimens should have received no more than 250mg mg/m2 prior to cisplatin.

Etoposide-Carboplatin Cohort:

• For dose levels 0-3, patients with untreated SCLC must have received two cycles of their first etoposide carboplatin regimen prior to registration to that chemotherapy cohort. For dose level 4, SCLC patients planned for the etoposide/carboplatin cohort may not have had prior chemotherapy regimens and do not have to have their first two cycles of etoposide-platinum prior to study entry.

Other Systemic Therapy:

* Patients may have received other prior therapies including immunotherapy, angiogenesis inhibitors, PARP inhibitors or signal transduction inhibitors. Patients who have received other treatment with PD-L1 / PD-1, CTLA4 or other antibodies must not have had intolerable toxicity or required steroids to manage toxicity.
* Patients must have recovered from all reversible toxicity related to prior chemotherapy or systemic therapy and have adequate washout as follows:

Longest of one of the following:

* Two weeks
* 5 half lives for investigational agents
* Standard cycle length of standard therapies

Radiation:

• Prior external beam radiation is permitted provided a minimum of 28 days (4 weeks) have elapsed between the last dose of radiation and date of registration. Exceptions may be made for low-dose, non-myelosuppressive radiotherapy after consultation with CCTG. Concurrent radiotherapy is not permitted. Patients planned for concurrent chemotherapy-radiation are not eligible. Patients with curative doses of radiation to marrow-bearing areas may not be eligible. Consult CCTG.

Surgery:

• Previous surgery is permitted provided that a minimum of 28 days (4 weeks) have elapsed between any major surgery and date of registration, and that wound healing has occurred.

* Patients must have recovered from any treatment related toxicities prior to registration (unless grade 1, irreversible, or considered by investigator as not clinically significant).
* Hematology:

Absolute neutrophils ≥ 1.5 x 10^9/L Platelets ≥ 100 x 10^9/L Hemoglobin ≥ 90 g/L

* Chemistry:

Bilirubin ≤ 1.5 x ULN (upper limit of normal) * If confirmed Gilbert's, eligible providing ≤ 3 x UNL; AST and ALT ≤ 2.5 x ULN (if liver metastases are present, ≤5 x UNL) Serum creatinine < 1.25 x ULN or: Creatinine clearance ≥ 50 mL/min

* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to registration in the trial and prior to tests which are considered to be study specific to document their willingness to participate.

Patients who cannot give informed consent (i.e. mentally incompetent patients, or those physically incapacitated such as comatose patients) are not to be recruited into the study. Patients competent but physically unable to sign the consent form may have the document signed by their nearest relative or legal guardian. Each patient will be provided with a full explanation of the study before consent is requested.

* Female patients of childbearing potential who are sexually active with a non sterilized male partner must use at least one highly effective method of contraception while on study and for 6 months after the last dose of durvalumab and tremelimumab or for 3 months after the last dose of durvalumab alone and consult product monograph for standard chemotherapy. Male partners of a female subject and non-sterilized male patients who are sexually active with a female partner of childbearing potential must use male condom plus spermicide while on study and for 6 months after the last dose of durvalumab and tremelimumab or for 3 months after the last dose of durvalumab alone and consult product monograph for standard chemotherapy. Female partners of a male subject must use a highly effective method of contraception throughout this period. Cessation of birth control after this point should be discussed with a responsible physician.
* Male patients should also refrain from donating sperm.
* Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial. Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, response assessment, adverse events, and follow-up.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient registration

Exclusion Criteria:

* Patients with a history of other malignancies requiring concurrent anticancer therapy.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease (e.g. colitis or Crohn's disease), diverticulitis with the exception of diverticulosis, celiac disease or other serious gastrointestinal chronic conditions associated with diarrhea), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis), rheumatoid arthritis, hypophysitis, uveitis, etc., within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

  * Patients with alopecia.
  * Patients with Grave's disease, vitiligo or psoriasis not requiring systemic treatment (within the last 2 years).
  * Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement.
* History of primary immunodeficiency, history of allogenic organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 28 days of registration* or a prior history of severe (grade 3 or 4) immune mediated toxicity from other immune therapy or grade ≥ 3 infusion reaction.

  * NOTE: Intranasal/inhaled corticosteroids or systemic steroids that do not to exceed 10 mg/day of prednisone or equivalent dose of an alternative corticosteroid are permissible.
* Live attenuated vaccination administered within 30 days prior to registration.
* History of hypersensitivity to durvalumab or tremelimumab or any excipient. Patients who have received other treatment with PD-L1 / PD-1, CTLA4 or other antibodies must not have had intolerable toxicity or required steroids to manage toxicity.
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 470 msec in screening ECG measured using standard institutional method or history of familial long QT syndrome.
* Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction within the previous year or cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects). Patients with a significant cardiac history, even if controlled, should have a LVEF ≥ 50%.
* Concurrent treatment with other investigational drugs or anti-cancer therapy.
* Patients with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol. This includes but is not limited to:

  * history of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements;
  * active infection requiring systemic therapy; (including any patient known to have active hepatitis B, hepatitis C or human immunodeficiency virus (HIV) or tuberculosis or any infection requiring systemic therapy);
  * active peptic ulcer disease or gastritis;
  * untreated symptomatic brain metastases or brain metastases in whom radiation or surgery is indicated.
  * pneumonitis
* Pregnant or lactating women. Women of childbearing potential must have a urine pregnancy test (urine or serum) proven negative within 14 days prior to registration.

Men and women of child-bearing potential must agree to use adequate contraception.

* Not able to receive the standard chemotherapy regimen (consult product monograph).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-10-16 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Confirm the recommended phase II dose (RP2D) of durvalumab ± tremelimumab in patients receiving standard chemotherapy | 24 months

SECONDARY OUTCOMES:
Number of Participants with treatment-related adverse events as assessed by CTCAE v 4.0 | 24 months
Efficacy of durvalumab ± tremelimumab in patients receiving standard chemotherapy. Assessed by chest/abdomen/pelvis CT scan and other scans as necessary to document | 24 months
  disease
Characterize the immunogenicity of durvalumab ± tremelimumab in patients receiving standard chemotherapy | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rosalyn Juergens, Study Chair — Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, ON Canada; Desiree Hao, Study Chair — Tom Baker Cancer Centre, Calgary, Alberta, Canada
Locations (7):
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Juergens RA, Hao D, Ellis PM, Tu D, Mates M, Kollmannsberger C, Bradbury PA, Tehfe M, Wheatley-Price P, Robinson A, Bebb G, Laskin J, Goffin J, Hilton J, Tomiak A, Hotte S, Goss GD, Brown-Walker P, Sun X, Tsao MS, Cabanero M, Gauthier I, Song X, Dennis PA, Seymour LK, Smoragiewicz M, Laurie SA. A phase IB study of durvalumab with or without tremelimumab and platinum-doublet chemotherapy in advanced solid tumours: Canadian Cancer Trials Group Study IND226. Lung Cancer. 2020 May;143:1-11. doi: 10.1016/j.lungcan.2020.02.016. Epub 2020 Feb 28. PMID 32169783